CLINICAL TRIAL: NCT02155634
Title: Phase 3b, Randomized Trial of Continuous Revlimid® (Lenalidomide) Therapy Versus Observation Following Induction Therapy That Does Not Include Revlimid, Pomalyst® or Thalomid® in Newly Diagnosed Multiple Myeloma
Brief Title: Continuous Lenalidomide Therapy Versus Observation Following Induction Without Lenalidomide, Pomalidomide or Thalidomide in Myeloma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to poor feasibility and lack of interest at the participating sites.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MM-027
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Multiple Myeloma; Neoplasms; Plasma Cells; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Therapeutic Uses
Keywords: Newly Diagnosed Multiple Myeloma; Multiple Myeloma; Lenalidomide; Revlimid; Phase III; Phase IIIb; Plasma Cell Dyscrasia
MeSH Terms: conditions — Multiple Myeloma; Neoplasms; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lenalidomide (Experimental): Lenalidomide maintenance given until disease progression. Long term follow-up 5 years post last patient randomized.
  Interventions: Drug: Lenalidomide
- Observation (No Intervention): Observation until disease progression. Long term follow-up 5 years post last patient randomized.

INTERVENTIONS:
Drug: Lenalidomide — Treatment with lenalidomide capsules 10 mg, 5mg daily or 5mg every other day given on days 1-21 of each 28 day cycle.
  Other Names: Revlimid
  Arms: Lenalidomide

SUMMARY:
The purpose of this study is to see how long lenalidomide therapy can maintain or improve the disease response obtained after induction therapy that does not include lenalidomide, pomalidomide or thalidomide; and consequently reduce worsening of disease and to evaluate the activity of lenalidomide. Patients will receive lenalidomide or be under observation. All patients will attend regular clinic visits to evaluate their disease and health. Patients will have the option to participate in additional biomarker correlative studies in addition to their participation in the main study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study: Related to initial diagnosis and prior induction

1. Previously untreated and symptomatic multiple myeloma (MM).
2. MM diagnosis meeting all 3 diagnostic criteria of (1) monoclonal plasma cells in the bone marrow ≥ 10% and/or presence of a biopsy-proven, plasmacytoma, (2) monoclonal protein in the serum and/or urine, and (3) at least one criteria of hypercalcemia, renal failure, anemia or bone disease.
3. Measurable disease by protein electrophoresis analyses.
4. All subjects must be treated with a minimum of 6 cycles (unless subject achieved a complete response prior to 6 cycles),and a maximum of 12 cycles of induction without lenalidomide (LEN), pomalidomide (POM) or thalidomide (THAL). Subject must have achieved at least stable disease (SD) as best overall response and maintained SD or better throughout the induction until screening. Subjects who plateau must have at least 2 cycles at best response prior to randomization.
5. Subjects must have cytogenetic (e.g.:17 p deletion, and 4;14 translocation), β-2 microglobulin and serum albumin (ISS Stage) results from their initial diagnosis available at the time of screening.

   Related to the subject
6. Must understand and voluntarily sign the informed consent document (ICD) prior to the conduct of any study related assessments/procedures,
7. Age ≥ 65 years: if < 65 years of age, the subject must be non eligible for or decline stem cell transplant,
8. Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2,
9. Able to adhere to the study visit schedules and other protocol requirements,
10. Females of Childbearing Potential * (FCBP) must:

    1. Have two negative pregnancy tests as verified by the study doctor prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after the end of study therapy. This applies even if the subject practices true abstinence** from heterosexual contact.
    2. Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis) or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting investigational product (IP), during the study therapy (including dose interruptions), and for 28 days after discontinuation of study therapy.
11. Male Subjects must:

    1. Practice true abstinence** or agree to use a condom during sexual contact with a pregnant female or a FCBP while participating in the study, during dose interruptions and for at least 28 days following IP discontinuation, even if he has undergone a successful vasectomy.
    2. Agree to not donate semen during IP therapy and for 28 days after end of study therapy.
12. All subjects must:

    1. Have an understanding that the study medication could have a potential teratogenic risk.
    2. Agree to abstain from donating blood while taking IP therapy and following discontinuation of IP therapy.
    3. Agree not to share study medication with another person.
    4. All FCBP and male subjects must be counseled about pregnancy precautions and risks of fetal exposure.

       * An FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (ie, amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).

         * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (et, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].

Exclusion Criteria:

* The presence of any of the following will exclude the subject from the study enrollment:

  1. Previous treatment with anti-myeloma therapy other than the required 6-12 cycles of induction without LEN, POM or THAL (does not include local radiotherapy, bisphosphonates, or a single short course of steroid [ie, less than or equal to the equivalent of dexamethasone 40 mg/day for 4 days; such a short course of steroid treatment must not have been given within 14 days of randomization]).
  2. Subjects who did not achieve SD or better after getting at least 6 cycles of induction are not eligible.
  3. Non-secretary MM.
  4. Prior therapy with LEN, POM, THAL or Melphalan. Subjects who received investigational agents are also excluded.
  5. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
  6. Pregnant or lactating females.
  7. Any of the following laboratory abnormalities:

     * Absolute Neutrophil Count (ANC) < 1,000/µL (1.0 x 109/L)
     * Untransfused platelet count < 50,000 cells/µL (50 x 109/L)
     * Serum aspartate aminotransferase (AST)/ serum glutamic oxaloacetic transaminase (SGOT) or alanine aminotransferase (ALT)/ serum glutamic pyruvic transaminase (SPGT) > 3.0 x upper limit of normal (ULN)
     * Serum bilirubin levels > 1.5 x ULN
  8. Severe renal insufficiency (creatinine clearance [CrCl] < 30 mL/min by Cockcroft-Gault method) or actual CrCl result requiring hemodialysis or peritoneal dialysis.
  9. Prior history of malignancies including skin cancer, other than multiple myeloma, with exception of basal cell carcinoma and squamous cell carcinoma in situ.
  10. Prior history of deep vein thrombosis or pulmonary embolism within 3 years of randomization.
  11. Subjects who are unable or unwilling to undergo anti-thrombotic therapy.
  12. Peripheral neuropathy of > Grade 2 severity according to the NCI CTCAE Version 4.0.
  13. Known Human immunodeficiency virus positivity or active infectious hepatitis, type A, B, or C.
  14. Primary amyloidosis (immunoglobulin light chain) and myeloma complicated by amyloidosis.
  15. Prior allogeneic or autologous stem cell transplantation.
  16. Significant active cardiac disease within the previous 6 months of signing the ICD including:

      * New York Heart Association class II-IV congestive heart failure
      * Unstable angina or angina requiring surgical or medical intervention
      * Myocardial infarction
  17. Any condition that confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2017-04 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Approximately 36 months.
  Time from randomization to the documentation of disease progression

SECONDARY OUTCOMES:
Response Rate | Approximately 36 months
  Response is defined according to the international Myeloma Working Group (IMWG) Response Criteria (Durie, 2006). Overall response rate over time (complete response [CR], very good partial response [VGPR], partial response [PR], stable disease [SD]
Time to progression (TTP) | Approximately 36 months
  The time to progression is defined from randomization to progression as defined by the international Myeloma Working Group (IMWG) Criteria (Durie, 2006)
Overall survival (OS) | Approximate 6.5 years
  Time from randomization to the date of death due to any cause
Safety | Approximate 6.5 years
  Number of patients with adverse events and relationship of adverse events, laboratory abnormalities, and hospitalizations to study drug / study observation

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Nagarwala, MD, Study Director — Celgene